CLINICAL TRIAL: NCT07336069
Title: The Research to Evaluate the Efficacy and Safety of the Shilangqing Smart Reading Aid for Improving Reading Ability in Children With Low Vision (SLQ-001)
Brief Title: Shilangqing Smart Reading Aid for Improving Reading Ability in Children With Low Vision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Yuan, PHD, Beijing Tongren Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022QXPJ001
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-07

CONDITIONS: Low Vision Aids

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Using the "Shilangqing" device, conduct reading practice at a brightness level of 400 nit, and measure the eye health indicators before and after the reading session.
  Interventions: Device: "Langshiqng" visual aid device

INTERVENTIONS:
Device: "Langshiqng" visual aid device — Using the "Langshiqng" visual aid device, conduct reading practice at a brightness level of 400 nit, and measure the eye health indicators before and after the reading session.

SUMMARY:
This clinical trial aims to assess the efficacy and safety of the Shilangqing Smart Reading Aid, a head-mounted device integrating XR and AI technologies, in improving reading performance and quality of life among children with low vision. The study employs a multicenter, randomized, controlled design with two parallel groups: an experimental group using the Shilangqing device and a control group using traditional optical magnifiers. Participants will undergo a 12-week intervention period, with primary outcomes focusing on reading speed, accuracy, and user satisfaction. Secondary outcomes include changes in visual acuity, eye health metrics (e.g., tear film stability, visual fatigue), and device-related adverse events. The trial builds on preliminary data from Zhongshan Ophthalmic Center and user feedback indicating high efficacy and safety. An estimated 120 participants aged 6-18 years with best-corrected visual acuity of 0.05 to <0.3 will be recruited from multiple sites in China. Results will inform clinical adoption and regulatory approvals for low-vision assistive devices.

ELIGIBILITY:
Inclusion Criteria:

* The study included healthy individuals older than 18 years of age with a best-corrected visual acuity (BCVA) of <0.1 logarithm of minimum angle of resolution (logMAR) and no ongoing or prior history of ocular or systemic disease.

Exclusion Criteria:

* The study excluded healthy individuals younger than 18 years of age with a best-corrected visual acuity (BCVA) of >0.1 logarithm of minimum angle of resolution (logMAR) with ongoing or prior history of ocular or systemic disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Asthenopia score | 30 min
  Participants completed the Visual Fatigue Subjective Scale questionnaire post 30-minute reading session (MEMC and non-MEMC). This 20-item scale assessed eye strain, headaches, perceived clarity, and general comfort, with responses analyzed to identify differences in subjective visual fatigue between conditions.

SECONDARY OUTCOMES:
Motion sickness score | 30 min
  Participants completed the Motion sickness Subjective Scale questionnaire post 30-minute reading session.
The first tear film break-up time | 30 min
  The first tear break-up time of the participants was measured using the ocular Surface Synthesis analyzer after the 30 min reading task
distance eye position | 30 min
  The distance eye position of the participants was measured using a Maddox rod after the 30-min reading task
near eye position | 30 min
  The near eye position of the participants was measured using a Maddox rod after the 30-min reading task
AC/A | 30 min
  AC/A of the participants was measured using Maddox rod after the 30-min reading task
Accommodative responses | 30 min
  Accommodative responses were measured using a comprehensive refractometer after the 30-min reading task
Intra-ocular pressure | 30 min
  Intra-ocular pressure were measured using a neural crest tumor after the 30-min reading task
visual acuity | 30 min
  The visual acuity of the participants were measured using the EDTRS visual acuity chart after the 30-min reading task

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Ophthalmology and Visual Sciences Key Laboratory, Beijing Tongren Eye Center, Beijing, China